CLINICAL TRIAL: NCT04708470
Title: A Phase I/II Study of Combination Immunotherapy for Advanced Cancers Including HPV-Associated Malignancies, Small Bowel, and Colon Cancers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210007; 21-C-0007
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12-19

CONDITIONS: Oropharyngeal Cancer; Neck Cancer; Human Papillomavirus; HPV; Anal Cancer; Cervical Cancer; Penile Cancer; Vulvar Cancer; Vaginal Cancer; Colon Cancer
Keywords: Bintrafusp Alfa M7824; Entinostat; PDS01ADC M9241; PD-1(L1); Immunotherapy
MeSH Terms: conditions — Oropharyngeal Neoplasms; Head and Neck Neoplasms; Anus Neoplasms; Uterine Cervical Neoplasms; Penile Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Colonic Neoplasms | interventions — bintrafusp alfa protein, human; entinostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/Arm 1 (Experimental): Dose escalation/de-escalation of entinostat and dose escalation of PDS01ADC with fixed dose of bintrafusp alfa
  Interventions: Drug: Bintrafusp Alfa; Drug: PDS01ADC; Drug: Entinostat
- 2/Arm 2 (Experimental): RP2D of entinostat, PDS01ADC, and bintrafusp alfa
  Interventions: Drug: Bintrafusp Alfa; Drug: PDS01ADC; Drug: Entinostat
- 3/Arm3 (Experimental): Entinostat and PDS01ADC (without bintrafusp alfa)
  Interventions: Drug: PDS01ADC; Drug: Entinostat

INTERVENTIONS:
Drug: Bintrafusp Alfa — Subjects will receive bintrafusp alfa via IV infusion over 1 hour (-10 minutes / +20 minutes, that is, over 50 to 80 minutes) once every 2 weeks. Bintrafusp alfa will be administered as a "flat" dose of 300 mg independent of body weight. Bintrafusp alfa is administered as an intravenous infusion with a mandatory 0.2 micron in-line filter.
  Arms: 1/Arm 1; 2/Arm 2
Drug: PDS01ADC — PDS01ADC will be administered at as dose of 4, 8, 12, or 16.8 micrograms/kg by SC injection every 2 or 4 weeks. The dose of PDS01ADC will be calculated based on the weight of the subject determined within 72 hours prior to the day of drug administration. The dose of PDS01ADC used for the previous administration can be repeated if the change in the subject's weight is 10% or less than the weight used for the last dose calculation.
Drug: Entinostat — The entinostat used in this study is a self-administered investigational agent and will be given orally at a designated dose once a week or as directed. Number of entinostat tablets will be calculated based on the dose for the participant.

SUMMARY:
Background:

Often, metastatic human papillomavirus (HPV) associated cancers cannot be cured. They also do not respond well to treatment. Some forms of colon cancer also have poor responses to treatment. Researchers want to see if a new drug treatment can help people with these types of cancers.

Objective:

To find a safe dose of entinostat in combination with PDS01ADC and bintrafusp alfa and to see if this treatment will cause tumors to shrink.

Eligibility:

Adults ages 18 and older who have cervical, oropharyngeal, anal, vulvar, vaginal, penile, squamous cell rectal, or another cancer that may be associated with HPV infection or microsatellite stable small bowel or colorectal cancer.

Design:

Participants will be screened with a medical history and physical exam. Their ability to do daily activities will be assessed. They may have imaging scans of the brain and/or chest, abdomen, and pelvis. They may have nuclear bone scans. They will have an electrocardiogram to test heart function. They will have blood and urine tests. They may have a tumor biopsy. Participants with skin lesions may have them photographed.

Some screening tests will be repeated during the study.

Treatment will be done in 28-day cycles. Participants will get bintrafusp alfa through an intravenous catheter every 2 weeks. They will get PDS01ADC as an injection under the skin every 4 weeks. They will take entinostat by mouth once a week. They will complete a medicine diary.

Participants will get treatment for 2 years. They will have 1-2 follow-up visits in the 30 days after treatment ends. Then they will be contacted every 6 months to check on their health.

DETAILED DESCRIPTION:
Background:

* Although PD-1(L1) inhibitors have been approved for the treatment of over a dozen different tumor types in recent years, the majority of patients with advanced cancer still do not respond to these agents, including patients with microsatellite stable (MSS) colon cancer and patients with checkpoint refractory cancers (e.g., oropharyngeal, cervical).
* Clinical studies suggest that treatment with a bifunctional fusion protein targeting PD-L1 and TGF beta (bintrafusp alfa) may help overcome resistance or refractoriness to anti PD-1(L1) therapy alone.
* Preclinical and clinical studies suggest that treatment with a histone deacetylase inhibitor (HDAC inhibitor) concomitantly with anti PD-1(L1) therapy is safe and may help overcome resistance or refractoriness to anti PD-1(L1) therapy alone.
* Preclinical and clinical studies suggest that treatment with a tumor targeted immunocytokine (PDS01ADC) concomitantly with anti PD-1(L1) therapy is safe and may help overcome resistance or refractoriness to anti PD-1(L1) therapy alone.
* Preclinical studies suggest that the use of a combination of multiple immunotherapy agents may have improved anti-tumor efficacy.

  * Specifically, preclinical studies have shown that the combination of three immunotherapy agents (1) an HDAC inhibitor, entinostat (2) a tumor targeted immunocytokine (PDS01ADC), and (3) a bifunctional fusion protein targeting PD-L1 and TGF beta (bintrafusp alfa) produces greater anti-tumor activity than single or dual combinations of these agents.

Objectives:

* Phase I: To determine the recommended phase II dose (RP2D) of entinostat in combination with PDS01ADC and bintrafusp alfa.
* Phase II: To evaluate the objective response rate (ORR) (PR+CR) according to Response Evaluation Criteria (RECIST 1.1) of the combination of entinostat, PDS01ADC, and bintrafusp alfa in two separate populations:

  * Checkpoint refractory human papillomavirus (HPV) associated malignancies;
  * MSS small bowel or colorectal cancer.

Eligibility:

* Age >= 18 years old.
* Phase I: Subjects with cytologically or histologically confirmed locally advanced or metastatic HPV associated malignancies or MSS small bowel or colorectal cancer (Cohort 1).
* Phase II: Subjects with cytologically or histologically confirmed locally advanced or metastatic HPV associated malignancies (Cohort 2), or MSS small bowel or colorectal cancer (Cohort 3).
* Prior first line systemic therapy is required unless the participant declines standard treatment after appropriate counseling has been provided.
* Subjects must have measurable disease per RECIST 1.1.

Design:

* This is a phase I/II trial of combination immunotherapy.
* Participants will be treated with a one week lead in of entinostat alone followed by the combination of entinostat, PDS01ADC and bintrafusp alfa (Arm 1 & Arm 2). Up to 12 additional participants will be treated with a one week lead in of entinostat alone followed by the combination with PDS01ADC (without bintrafusp alfa, Arm 3).
* Phase I (Arm 1):

  * Arm 1 will be conducted using dose escalation/de-escalation of entinostat and dose escalation of PDS01ADC with a fixed dose of bintrafusp alfa in Cohort 1 (up to 36 total).
  * Once the combination of all three agents has been determined to be safe, participants from Cohort 2 and Cohort 3 may enroll into -Phase II.
* Phase II (Arm 2 and Arm 3):

  * (Arm 2) will be conducted using a Simon optimal two-stage design.
  * Cohort 2 (checkpoint refractory HPV associated malignancies, 16 total) and cohort 3 (MSS small bowel or colorectal cancer, 16 total) participants will each be enrolled to Arm 2.
  * If one or more out of twelve participants in a given cohort (2 or 3) has an objective response, accrual will be expanded to enroll 16 evaluable participants on that cohort.
  * If 3 or more of 16 (18.8%) participants respond in a given cohort-arm combination, that would be sufficiently interesting to warrant further study of the combination in later trials in that disease type.
  * Arm 3: Up to 12 additional participants with checkpoint refractory HPV associated cancer may enroll to the combination of entinostat plus PDS01ADC (without bintrafusp alfa).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Phase I: Subjects with cytologically or histologically confirmed locally advanced or metastatic HPV associated malignancies or MSS small bowel or colorectal cancer (Cohort 1).
* Phase II: Subjects with cytologically or histologically confirmed locally advanced or metastatic HPV associated malignancies (Cohort 2), or MSS small bowel or colorectal cancer (Cohort 3).
* Cohort 2 includes:

  * Cervical cancers;
  * P16+ Oropharyngeal cancers;
  * Anal cancers;
  * Vulvar, vaginal, penile, and squamous cell rectal cancers;
  * Other locally advanced or metastatic solid tumors (e.g., lung, esophagus) that are known HPV+.
* Subjects with MSS colorectal or small bowel cancer must have received two prior lines of systemic chemotherapy. Subjects with HPV associated malignancies must have received one prior line of systemic chemotherapy as well as checkpoint therapy if checkpoint therapy is FDA approved for that specific tumor type (e.g., HNSCC and PDL1+ cervical cancer). Prior checkpoint therapy is not needed where checkpoint therapy has not been FDA approved for that specific tumor type (e.g., anal, vaginal, vulvar, penile, PDL1 negative cervical). Exceptions to the above include participant who are not eligible to receive the above therapies or who decline these standard treatment options after appropriate counseling has been provided.
* Subjects must have measurable disease, per RECIST 1.1.
* Age >=18 years.
* ECOG performance status <=2
* Adequate hematologic function at screening, as follows:

  * Absolute neutrophil count (ANC) >=1.5 x 10^9/L;
  * Hemoglobin >= 9 g/dL;
  * Platelets >= 100,000/microliter.
* Adequate renal and hepatic function at screening, as follows:

  * Measured or calculated creatinine clearance (using the Cockcroft-Gault equation) > 50 mL/min
  * Bilirubin <= 1.5 x ULN OR in subjects with Gilbert s syndrome, a total bilirubin <= 3.0 x ULN
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2.5 x ULN, unless liver metastases are present, then values must be <= 3 x ULN).
* The effects of the immunotherapies on the developing human fetus are unknown. For this reason and because immunotherapeutic agents as well as other therapeutic agents used in this trial are known to be teratogenic, individuals of child-bearing potential and those who can father children must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) at the study entry and for 4 months after the last bintrafusp alfa dose, 3 months after the last entinostat dose and 2 months after the last PDS01ADC dose, whichever occurs later.
* Participants serologically positive for HIV, Hep B, Hep C are eligible as long as the viral loads are undetectable by quantitative PCR. HIV positive participants must have CD4 count >= 200 cells per cubic millimeter at enrollment, be on stable antiretroviral therapy for at least 4 weeks and have no reported opportunistic infections or Castleman's disease within 12 months prior to enrollment.
* Subjects must be able to understand and be willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants with prior investigational drug, chemotherapy, immunotherapy or any prior radiotherapy (except for palliative bone directed therapy) within the past 28 days prior to enrollment except if the investigator has assessed that all residual treatment-related toxicities have resolved or are at grade 1 severity and feel the participant is otherwise suitable for enrollment.
* Administration of live vaccine within 30 days prior to enrollment
* Major surgery within 28 days prior to enrollment (minimally invasive procedures such as diagnostic biopsies are permitted).
* Known active brain or central nervous system metastasis (less than a month out from definitive radiotherapy or surgery), seizures requiring anticonvulsant treatment (<3 months) or clinically significant cerebrovascular accident (<3 months). In order to be eligible participants must have repeat CNS imaging at least a month after definitive treatment showing CNS disease that has not progressed. Participants with CNS disease that has not progressed at least a month after definitive treatment and continued on <=10 mg of prednisone (or equivalent) for treatment of brain or central nervous system metastasis are eligible to enroll in this study. Participants with evidence of intratumoral or peritumoral hemorrhage on baseline imaging are also excluded unless the hemorrhage is grade <= 1 and has been shown to be stable on two consecutive imaging scans.
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with exception of:

  * Diabetes type I, eczema, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease or other mild autoimmune disorders not requiring immunosuppressive treatment;
  * Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable;
* Subjects on systemic intravenous or oral corticosteroid therapy with the exception of hormone replacement or physiologic doses of corticosteroids (<= the equivalent of prednisone 10 mg/day) or other immunosuppressive drugs such as azathioprine or cyclosporin A are excluded on the basis of potential immune suppression. For these subjects these excluded treatments must be discontinued at least 1 weeks prior to enrollment for recent short course use (<= 14 days) or discontinued at least 4 weeks prior to enrollment for long term use (> 14 days). In addition, the use of corticosteroids as premedication for contrast-enhanced studies is allowed prior to enrollment and on study.
* Subjects with a history of serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, bleeding diathesis or recent (within 3 months before enrollment) clinically significant bleeding events, or other illness or medical condition considered by the Investigator as high risk for investigational drug treatment. Note: For participants otherwise eligible to be assigned to receive just PDS01ADC and entinostat (without bintrafusp alfa, Arm 3), bleeding diathesis or recent bleeding will not be an exclusion.
* Subjects unwilling to accept blood products as medically indicated.
* Subjects with conditions associated with significant necrosis of nontumor-bearing tissues: esophageal or gastroduodenal ulcers < 3 months prior to enrollment, organ infarction < 3 months prior to enrollment, or active ischemic bowel disease.
* Presence of medically significant third space fluid (symptomatic pericardial effusion, ascites or pleural effusion requiring repetitive paracentesis).
* History of second malignancy within 3 years of enrollment except for the following: adequately treated localized skin cancer, cervical carcinoma in situ, superficial bladder cancer, or other localized malignancy which has been adequately treated or malignancy

which does not require active systemic treatment (e.g. low risk chronic lymphocytic leukemia (CLL)).

* Subjects with a known severe hypersensitivity reaction to compounds of similar chemical or biologic composition to any of study drugs (grade >/= 3 NCI-CTCAE v5) will be evaluated by the allergy/immunology team prior to enrollment.
* Pregnant individuals are excluded from this study because these drugs have not been tested in pregnant individuals and there is potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these immunotherapies, nursing should be discontinued if the mother is treated on this protocol.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Ojective response rate (ORR) of triple combination | two years
  Phase II: To evaluate the objective response rate (ORR) according to Response Evaluation Criteria (RECIST 1.1) of the combination of entinostat, PDS01ADC, and bintrafusp alfa in two separate populations: checkpoint refractory HPV associated malignancies and MSS small bowel or colorectal cancer
Determine RP2D of entinostat | two years
  Phase I: To determine the recommended phase II dose (RP2D) of entinostat in combination with PDS01ADC and bintrafusp alfa

SECONDARY OUTCOMES:
Safety of Triple Combination Therapy | two years
  Phase II: To evaluate the safety of the combination of entinostat, PDS01ADC, and bintrafusp alfa in subjects with advanced malignancies
Progression-Free Survival (PFS) | two years
  Phase II: To assess progression-free survival (PFS), and duration of response (DoR) for each population (HPV, Colon) according to RECIST 1.1.
Hospitalization due to AEs attributed to PD | two years
  Phase II: To assess proportion of participants that are hospitalized because of adverse events attributed to disease progression.
Duration of Response (DoR) | two years
  Phase II: To assess progression-free survival (PFS), and duration of response (DoR) for each population (HPV, Colon) according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Hoyoung M Maeng, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2021-C-0007.html